CLINICAL TRIAL: NCT07299513
Title: Aerodigestive Fistulas in Adults: Management at the Strasbourg University Hospital Between 2014 and 2023
Brief Title: Aerodigestive Fistulas in Adults at the University Hospital of Strasbourg
Acronym: FAD'HUS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9376
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Aerodigestive Fistulas
Keywords: Aerodigestive fistulas; Endoscopic investigations; Thoracic cancer; Oncological disease; Malignant fistula

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acquired aerodigestive fistulas in adults are rare conditions, corresponding to a pathological communication between the digestive and respiratory tracts, requiring collaborative multidisciplinary management. Clinical manifestations are nonspecific, ranging from a simple cough to pulmonary sepsis, which can be life-threatening. Diagnosis is often multimodal, requiring radiological examinations and endoscopic investigations. The most frequent etiologies are divided into two groups: benign and malignant causes, each group representing 50% of all acquired aerodigestive fistulas. Among the benign etiologies, 75% are iatrogenic, mainly represented by complications related to orotracheal intubation. These fistulas of benign etiology most often have a favorable prognosis, amenable to surgical treatment. Conversely, the development of an aerodigestive fistula in the context of thoracic cancer marks a turning point in the evolution of the oncological disease. Indeed, the average life expectancy of patients with a malignant fistula is estimated at between 1 and 6 weeks without specific treatment. Following this palliative approach aimed at improving quality of life, multiple treatment options are available, often combined with digestive and thoracic endoscopy.

The Strasbourg University Hospitals are a leading tertiary care center for these pathologies, with departments of Pulmonology, Gastroenterology, Digestive Surgery, Thoracic Surgery, Medical Intensive Care, Multipurpose Surgical Intensive Care, Bronchial Endoscopy, and Digestive Endoscopy. The centre's influence extends over the entire eastern part of the Grand Est region (Nancy, Metz, Strasbourg, Mulhouse).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years at diagnosis
* Diagnosis between January 1, 2014, and December 31, 2023
* Aerodigestive fistula defined by one of the following criteria:
* Fistula visualized by bronchoscopy and/or digestive endoscopy
* Fistula visualized by static chest imaging (CT scan or MRI)
* Fistula visualized by dynamic chest imaging (barium swallow)
* Hospitalization at the Strasbourg University Hospitals (HUS)

Exclusion Criteria:

* Explicit refusal by the patient to provide their data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult subject with a fAerodigestive fistula between January 1, 2014, and December 31, 2023
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11-21 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate since diagnosis | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pneumologie - Hôpitaux Universitaires de Strasbourg, Strasbourg, France